CLINICAL TRIAL: NCT04627818
Title: Diagnostic, Therapeutic and Reproductive Aspects of Patients with Mullerian Anomalies: a Prospective Cohort
Brief Title: Diagnostic, Therapeutic and Reproductive Aspects of Patients with Mullerian Anomalies
Acronym: MULAN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B6702020000011
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mullerian Anomaly of Uterus, Nec; Mullerian Anomaly of Vagina; Mullerian Anomaly of Cervix
Keywords: Mullerian anomaly; Diagnostic tools; Surgical treatment; Reproductive function; Obstetric complications
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with a mullerian variation

SUMMARY:
The purpose of this study is to get a better understanding of the clinical implications (including reproductive problems and obstetric complications), appropriate diagnostic tools and correct surgical treatment of Mullerian anomalies.

DETAILED DESCRIPTION:
Mullerian anomalies are rare, therefore they are not well known and not often considered as differential diagnosis. This causes a delay in the diagnosis with risk of long lasting symptoms and adverse effects on the reproductive function. However, the diagnosis can be made more accurately with improved diagnostic tools. Moreover, minimally invasive surgery allows for preservation and potential improvement of fertility in these women.

The purpose of this study is to get a better understanding of the clinical implications (including reproductive problems and obstetric complications), appropriate diagnostic tools and correct surgical treatment of Mullerian anomalies.

ELIGIBILITY:
Inclusion Criteria:

* women with a uterus
* presence of a mullerian variation
* Maximum age 45y

Exclusion Criteria:

* women without a uterus
* aged >45y

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — women with a uterus
Study Population: diagnosed and/or treated in the Ghent University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Fertility | 10 years after trying to conceive
  Time to clinical pregnancy
Fertility | 18 weeks after conception
  Early pregnancy loss
Surgical approach | During surgery
  Different surgical approaches used
Surgical success | 15 years after surgery
  Relief of symptoms after surgery

SECONDARY OUTCOMES:
Diagnostic accuracy | at the time of diagnostic workup
  The ability of a test to detect a Mullerian variation when it is present and detect the absence of a Mullerian variation when it is absent
Obstetric complications | 1 year after conception
  Complications during pregnancy, labor, delivery, and the postpartum period

CONTACTS AND LOCATIONS:
Overall Officials: Tjalina Hamerlynck, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided